CLINICAL TRIAL: NCT06774885
Title: ROLE OF FOLIC ACID IN THE MANAGEMENT OF ADJUVANT ENDOCRINE THERAPY-INDUCED HOT FLASHES IN BREAST CANCER PATIENTS
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Fatma Abdalkarim, Teaching Assistant- Pharmacy Practice & Clinical Pharmacy, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15/2025
Record Dates: First submitted 2025-01-09; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: THERAPY-INDUCED HOT FLASHES IN BREAST CANCER PATIENTS
Keywords: Breast cancer; Hot flashes; Endocrine therapy; Folic acid
MeSH Terms: conditions — Breast Neoplasms; Hot Flashes | interventions — Folic Acid; Tablets

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): The patient will not be administered with any drug/placebo
- Intervention (Experimental): 1mg of folic acid
  Interventions: Drug: Folic Acid 1 Mg Oral Tablet
- Treatment (Experimental): 5mg of folic acid
  Interventions: Drug: Folic Acid 5 Mg Oral Tablet

INTERVENTIONS:
Drug: Folic Acid 1 Mg Oral Tablet — 1 mg oral folic acid tablet
  Arms: Intervention
Drug: Folic Acid 5 Mg Oral Tablet — 5 mg oral folic acid tablet
  Arms: Treatment

SUMMARY:
The study's objective is to investigate the role of folic acid administration in the management of hot flashes associated with adjuvant endocrine therapy in patients with breast cancer.

DETAILED DESCRIPTION:
Folic acid is one of the B vitamins that when absorbed into its active form is converted to tetrahydrofolate. Folate is an essential cofactor for the biosynthesis of norepinephrine and serotonin. Studies have also noted that folate, with a mechanism like hormone replacement therapy (HRT), can improve hot flashes by interfering with monoamine neurotransmitters called norepinephrine and serotonin .The purpose of the current study is to investigate the role of folic acid administration in the management of hot flashes associated with adjuvant endocrine therapy in patients with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Females older than 18 years
* Diagnosed with confirmed breast cancer and currently treated with an adjuvant endocrine
* Experiencing bothersome hot flashes at least 14 times/week
* Taking the treatment within 6 months to two years.

Exclusion Criteria:

* Known hypersensitivity to folic acid
* Patients who have been treated with selective serotonin reuptake inhibitors (SSRIs) within the past 30 days.
* Renal impairment is defined as a serum creatinine level greater than 2 mg/ld..
* Significant liver disease: Indicated by liver enzyme levels exceeding two times the upper limit of normal.
* Metastatic breast cancer
* Taking other medication for hot flashes
* Medications inducing hot flashes such as (Clomiphene, Opioids, Nifedipine, Prednisone)

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-02-09 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Reduction in Hot Flash Frequency and Severity | 3 months
  It is measured using the daily hot flash diary, which tracks the number and intensity of hot flashes over the study period.

SECONDARY OUTCOMES:
Improvement in Quality of Life | 3 months
  Assessed through the Hot Flash Related Daily Interference Scale (HFRDIS), which evaluates how hot flashes interfere with daily activities and overall well-being.
Correlation with Folic Acid Blood Levels | 3 months
  Folic acid levels in the blood will be measured to explore the relationship between serum folate concentrations and changes in hot flashes symptoms.

IPD SHARING:
Plan to Share IPD: No